CLINICAL TRIAL: NCT07170657
Title: Teen Recovery Through Inspiration, Support, and Empowerment (RISE)
Brief Title: Teen Recovery Through Inspiration, Support, and Empowerment
Acronym: Teen RISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Guillory, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2024-0493
Record Dates: First submitted 2025-08-11; First posted 2025-09-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Suicidal Ideation; Suicide Attempt; Anxiety; Depression Disorders
Keywords: Peer Support Specialist (PSS); Recovery Education and Support (RES) Program; Teenage; High School Teen; UT Southwestern Medical Center; Mental Health Recovery; Online; Virtual
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Cohort A: Intervention Group Cohort B: Standard of Care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: Intervention Group with PSS, TP, and RES (Experimental): Virtual one on one meetings peer support specialist (PSS), trained peer (TP) using recovery education and support program (RES). Group meetings with PSS, TP, and other participants. Qualitative and quantitative assessments.
  Interventions: Behavioral: Peer Support Services Recovery
- Cohort B: Standard of Care (No Intervention): Scheduled telephone call visit with a member of the research team. Qualitative and quantitative assessments.

INTERVENTIONS:
Behavioral: Peer Support Services Recovery — A program of mental health recovery through one-on-one and small group meetings with a PSS and TP using RES for individuals recently discharged from an acute care psychiatric facility.
  Arms: Cohort A: Intervention Group with PSS, TP, and RES

SUMMARY:
The goal of this pilot study is to test the effectiveness of a novel intervention for teenagers (ages 15-18) with mental health conditions who have been released from an acute care psychiatric facility. The intervention aims to reduce suicidality, depression, anxiety, re-hospitalization, and to improve mental health recovery by using an online recovery education and support program.

The current standard of care (SOC) for these patients at discharge includes a discharge plan with a list of their medication(s), anticipated outpatient appointment(s), and corresponding information on when and where to find community resources.

The intervention being tested involves the implementation of an online recovery education and support (RES) program, involving one-on-one and small group meetings led by trained teen peers (TPs) and peer support specialists (PSS).

Participants will be assigned to either Cohort A or B for 8 weeks.

Cohort A will be the intervention group with online access to an RES, TP, and PSS.

* Week 1-4: One-on-one meetings with PSS and TP for education and support. Assessments will be completed at week 2 and 4.
* Week 5 and 7: one-one meetings with PSS and TP for education and support.
* Week 6 and 8: small group meetings with PSS, TP, and other participants. Assessments will be completed during Weeks 6 and 8.

Cohort B will be the SOC group with no PSS, TP, or RES.

* Weeks 1-4: Weekly check in phone calls with a member of the research team. Assessments will be completed at Weeks 2 and 4.
* Weeks 5-8: Check in phone calls with a member of the research team every other week. Assessments will be completed at weeks 6 and8.

Data collected from participant assessments, adherence to medication, and re-admittance to a psychiatric facility will be used to compare the intervention to the SOC.

DETAILED DESCRIPTION:
Purpose:

* This is a pilot study to test the effectiveness of a novel intervention aimed at reducing the incidences of suicidality, depression, anxiety, re-hospitalization rates, and improving mental health recovery by utilizing outpatient services, and medication adherence for high school teenagers ages 15-18, with mental health conditions verses the standard of care (SOC) at discharge which only provides a discharge plan with a list of their medication(s), anticipated outpatient appointment(s), and corresponding information on when and where to find community resources.
* The intervention will use trained peers (TP), peer support specialists (PSS), and an online recovery education and support (RES) platform aimed at improving knowledge, awareness, and utilization of recovery and wellness programs for those patients recently discharged from an acute psychiatric treatment facility.

Objectives:

* Implement a program of mental health recovery education and support through virtual one-on-one and small group meetings with a TP and PSS for individuals recently discharged from an acute care psychiatric facility to determine the effectiveness of: Reduction of suicidality, depression, anxiety, re-hospitalization rate AND Improvement in mental health recovery by participating in outpatient services, and medication adherence.
* Determine if peer-led interventions improve knowledge, awareness, and utilization of recovery and wellness programs and support.

Endpoints:

* Determine the efficacy of peer-led, virtual one-on-one and group sessions vs standard of care (SOC) based on responses to assessments, adherence to medication, and re-admittance to a psychiatric facility.
* Determine if there is a difference in outcome based on demographics (race, ethnic background, diagnosis, public vs private insurance, and zip code)

Study Design:

- This is a 1:1 randomized, 8-week interventional study that will include an orientation session and a collection of baseline data. At the conclusion of the orientation session, subjects will be randomly assigned to Cohort A or B. Target recruitment is 40 for this study; 20 subjects in Cohort A and 20 in Cohort B. At the conclusion of the study, both groups will be provided a list resources for therapy, outpatient psychiatry providers/services, online recovery education and support (RES), local emergency departments and inpatient psychiatric facilities.

Cohort A - Intervention group with RES, PSS, and TP

* Weeks 1-4: one-on-one meetings with peer support specialist (PSS) for education and support. Qualitative and quantitative assessments completed at weeks 2 and 4
* Weeks 5-8: Biweekly (every other week) of one-on-one meetings with PSS and TP for education and support. Biweekly group meetings with PSS, TP, and other participants. Qualitative and quantitative assessments completed at weeks 6 and 8

Cohort B - SOC group with no PSS, TP, or RES; participants are responsible for finding resources or group support by following the information provided at discharge

* Weeks 1-4: Weekly check-in phone calls with a member of the research team. Qualitative and quantitative assessments completed at weeks 2 and 4 (completed during phone call check in)
* Weeks 5-8: Biweekly (every other week) check-in phone calls with a member of the research team. Qualitative and quantitative assessments completed at weeks 6 and 8 (completed during phone call check in).

ELIGIBILITY:
Inclusion Criteria:

* Chief complaint of suicidal ideation, suicide attempt, depression, and/or anxiety
* recently discharged from inpatient care or from emergency department
* men and women ages 15-18 years old

Exclusion Criteria:

- primary diagnosis of: substance use disorder, schizophrenia spectrum, intellectual development disorder, autism spectrum disorder (level II or III)

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in Suicidal Ideation as measured by C-SSRS at 2 weeks from baseline | Baseline, 2 weeks
  Change in suicidal ideation is measured by Columbia Suicide Severity Rating Scale (C-SSRS) at 2 weeks from baseline using both the baseline and since last visit assessment versions. Scoring of the assessment indicates severity. The C-SSRS consists of 16 questions that ask about suicidal ideation and behaviors (the first 10 questions comprise the ideation subscale and the last 6 comprise the behavior subscale). Total score ranges for suicidal ideation from a minimum of 0 (corresponding to no suicidal ideation) to a maximum of 5 (representing active suicidal ideation with plan and intent). Total score ranges for suicidal behavior from a minimum of 0 (corresponding to no suicidal behavior) to a maximum of 5 (representing active suicidal behavior).
Change in Suicidal Ideation as measured by C-SSRS at 4 weeks from baseline | Baseline, 4 weeks
  Change in suicidal ideation is measured by Columbia Suicide Severity Rating Scale (C-SSRS) at 4 weeks from baseline using both the baseline and since last visit assessment versions. Scoring of the assessment indicates severity. The C-SSRS consists of 16 questions that ask about suicidal ideation and behaviors (the first 10 questions comprise the ideation subscale and the last 6 comprise the behavior subscale). Total score ranges for suicidal ideation from a minimum of 0 (corresponding to no suicidal ideation) to a maximum of 5 (representing active suicidal ideation with plan and intent). Total score ranges for suicidal behavior from a minimum of 0 (corresponding to no suicidal behavior) to a maximum of 5 (representing active suicidal behavior).
Change in Suicidal Ideation as measured by C-SSRS at 6 weeks from baseline | Baseline, 6 weeks
  Change in suicidal ideation is measured by Columbia Suicide Severity Rating Scale (C-SSRS) at 6 weeks from baseline using both the baseline and since last visit assessment versions. Scoring of the assessment indicates severity. The C-SSRS consists of 16 questions that ask about suicidal ideation and behaviors (the first 10 questions comprise the ideation subscale and the last 6 comprise the behavior subscale). Total score ranges for suicidal ideation from a minimum of 0 (corresponding to no suicidal ideation) to a maximum of 5 (representing active suicidal ideation with plan and intent). Total score ranges for suicidal behavior from a minimum of 0 (corresponding to no suicidal behavior) to a maximum of 5 (representing active suicidal behavior).
Change in Suicidal Ideation as measured by C-SSRS at 8 weeks from baseline | Baseline, 8 weeks
  Change in suicidal ideation is measured by Columbia Suicide Severity Rating Scale (C-SSRS) at 8 weeks from baseline using both the baseline and since last visit assessment versions. Scoring of the assessment indicates severity. The C-SSRS consists of 16 questions that ask about suicidal ideation and behaviors (the first 10 questions comprise the ideation subscale and the last 6 comprise the behavior subscale). Total score ranges for suicidal ideation from a minimum of 0 (corresponding to no suicidal ideation) to a maximum of 5 (representing active suicidal ideation with plan and intent). Total score ranges for suicidal behavior from a minimum of 0 (corresponding to no suicidal behavior) to a maximum of 5 (representing active suicidal behavior).

SECONDARY OUTCOMES:
Changes in symptoms associated with anxiety as measured by GAD 7 at 2 weeks | Baseline, 2 weeks
  A reduction of anxiety symptoms and rates of occurrence will be measured using the Generalized Anxiety Disorder (GAD) 7 - a widely used screening tool for assessing the severity of generalized anxiety disorder (GAD) and consists of 7 items that evaluate anxiety symptoms with 4 response options: 0- "Not at all", 1-"Several days", 2-"More than half the days", 3-"Nearly every day". Total score can range from 0 to 21 with higher scores indicating higher levels of anxiety.
Changes in symptoms associated with anxiety as measured by GAD 7 at 4 weeks | Baseline, 4 weeks
  A reduction of anxiety symptoms and rates of occurrence will be measured using the Generalized Anxiety Disorder (GAD) 7 - a widely used screening tool for assessing the severity of generalized anxiety disorder (GAD) and consists of 7 items that evaluate anxiety symptoms with 4 response options: 0- "Not at all", 1-"Several days", 2-"More than half the days", 3-"Nearly every day". Total score can range from 0 to 21 with higher scores indicating higher levels of anxiety.
Changes in symptoms associated with anxiety as measured by GAD 7 at 6 weeks | Baseline, 6 weeks
  A reduction of anxiety symptoms and rates of occurrence will be measured using the Generalized Anxiety Disorder (GAD) 7 - a widely used screening tool for assessing the severity of generalized anxiety disorder (GAD) and consists of 7 items that evaluate anxiety symptoms with 4 response options: 0- "Not at all", 1-"Several days", 2-"More than half the days", 3-"Nearly every day". Total score can range from 0 to 21 with higher scores indicating higher levels of anxiety.
Changes in symptoms associated with anxiety as measured by GAD 7 at 8 weeks | Baseline, 8 weeks
  A reduction of anxiety symptoms and rates of occurrence will be measured using the Generalized Anxiety Disorder (GAD) 7 - a widely used screening tool for assessing the severity of generalized anxiety disorder (GAD) and consists of 7 items that evaluate anxiety symptoms with 4 response options: 0- "Not at all", 1-"Several days", 2-"More than half the days", 3-"Nearly every day". Total score can range from 0 to 21 with higher scores indicating higher levels of anxiety.
Changes in symptoms associated with depression as measured by PHQ-9 at 2 weeks | Baseline, 2 weeks
  A reduction of depression symptoms and rates of occurrence will be measured using the Patient Health Questionnaire (PHQ) - a self reported inventory used as a screening and diagnostic tool for depression.
  The PHQ-9 is a 9-item self-reported instrument that measures depression symptoms. Respondents are asked how much each symptom has bothered them over the past 2 weeks, with response options of "not at all", "several days", "more than half the days", and "nearly every day", scored as 0, 1, 2, and 3. The scale can range from 0 to 27, with higher scores indicating higher levels of depression.
Changes in symptoms associated with depression as measured by PHQ-9 at 4 weeks | Baseline, 4 weeks
  A reduction of depression symptoms and rates of occurrence will be measured using the Patient Health Questionnaire (PHQ) - a self reported inventory used as a screening and diagnostic tool for depression.
  The PHQ-9 is a 9-item self-reported instrument that measures depression symptoms. Respondents are asked how much each symptom has bothered them over the past 2 weeks, with response options of "not at all", "several days", "more than half the days", and "nearly every day", scored as 0, 1, 2, and 3. The scale can range from 0 to 27, with higher scores indicating higher levels of depression.
Changes in symptoms associated with depression as measured by PHQ-9 at 6 weeks | Baseline, 6 weeks
  A reduction of depression symptoms and rates of occurrence will be measured using the Patient Health Questionnaire (PHQ) - a self reported inventory used as a screening and diagnostic tool for depression.
  The PHQ-9 is a 9-item self-reported instrument that measures depression symptoms. Respondents are asked how much each symptom has bothered them over the past 2 weeks, with response options of "not at all", "several days", "more than half the days", and "nearly every day", scored as 0, 1, 2, and 3. The scale can range from 0 to 27, with higher scores indicating higher levels of depression.
Changes in symptoms associated with depression as measured by PHQ-9 at 8 weeks | Baseline, 8 weeks
  A reduction of depression symptoms and rates of occurrence will be measured using the Patient Health Questionnaire (PHQ) - a self reported inventory used as a screening and diagnostic tool for depression.
  The PHQ-9 is a 9-item self-reported instrument that measures depression symptoms. Respondents are asked how much each symptom has bothered them over the past 2 weeks, with response options of "not at all", "several days", "more than half the days", and "nearly every day", scored as 0, 1, 2, and 3. The scale can range from 0 to 27, with higher scores indicating higher levels of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Guillory, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
At this time - there is no intention of sharing individual participant data as this is a pilot study, and due to the relatively small number of participants, any data that is shared or published will be in aggregate.

REFERENCES:
- [Background] Peer Support Services. Texas Health and Human Services. (2019). Retrieved February 21, 2023, from https://www.hhs.texas.gov/providers/behavioral-health-services-providers/peer-support-services.
- [Background] White S, Foster R, Marks J, Morshead R, Goldsmith L, Barlow S, Sin J, Gillard S. The effectiveness of one-to-one peer support in mental health services: a systematic review and meta-analysis. BMC Psychiatry. 2020 Nov 11;20(1):534. doi: 10.1186/s12888-020-02923-3. PMID 33176729
- [Background] Lyons N, Cooper C, Lloyd-Evans B. A systematic review and meta-analysis of group peer support interventions for people experiencing mental health conditions. BMC Psychiatry. 2021 Jun 23;21(1):315. doi: 10.1186/s12888-021-03321-z. PMID 34162340
- [Background] Walker G, Bryant W. Peer support in adult mental health services: a metasynthesis of qualitative findings. Psychiatr Rehabil J. 2013 Mar;36(1):28-34. doi: 10.1037/h0094744. PMID 23477647
- [Background] Davidson L, Bellamy C, Guy K, Miller R. Peer support among persons with severe mental illnesses: a review of evidence and experience. World Psychiatry. 2012 Jun;11(2):123-8. doi: 10.1016/j.wpsyc.2012.05.009. PMID 22654945
- [Background] Nugent C. SAMSHA's working definition of recovery. In: SAMSHA, editor. 2012. p. 8.
- [Background] Soe K, Babajide A, Gibbs T (2019). American Psychiatric Association Position Statement on Transitional Age Youth. American Psychiatric Association. Accessed from https://www.psychiatry.org/home/policy-finder?k=adolescent
- [Background] Centers for Disease Control and Prevention. (2022). Web-based Injury Statistics Query and Reporting System (WISQARS). Atlanta, GA: National Centers for Injury Prevention and Control, Centers for Disease Control and Prevention. Retrieved from https://www.cdc.gov/injury/wisqars/index.html.
- [Background] Merikangas KR, He JP, Burstein M, Swanson SA, Avenevoli S, Cui L, Benjet C, Georgiades K, Swendsen J. Lifetime prevalence of mental disorders in U.S. adolescents: results from the National Comorbidity Survey Replication--Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry. 2010 Oct;49(10):980-9. doi: 10.1016/j.jaac.2010.05.017. Epub 2010 Jul 31. PMID 20855043
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837